CLINICAL TRIAL: NCT07370038
Title: Implementing the Unified Protocol for Burnout (UP-B): A Feasibility and Acceptability Study.
Brief Title: Feasibility and Acceptability of the Unified Protocol for Burnout
Acronym: UP-B
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F&A:UP-B
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Clinical Burnout
Keywords: transdiagnostic; cognitive-behavioral intervention; clinical burnout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unified Protocol for Burnout (Experimental): All participants will be included in this program.
  Interventions: Behavioral: Unified Protocol for Burnout

INTERVENTIONS:
Behavioral: Unified Protocol for Burnout — During the intervention, participants will complete eight modules designed to equip them with a defined set of skills for managing clinical burnout (i.e., understanding emotions, mindful emotion awareness, awareness and confrontation of physical sensations, cognitive flexibility, enhancement of cognitive functioning, and emotion-focused exposures). After each module, participants will be assigned homework exercises, which will be reviewed and discussed during the subsequent session.

SUMMARY:
The present study has three primary objectives: (1) to evaluate the feasibility of implementing the Unified Protocol for Burnout (UP-B) an intervention derived from the Unified Protocol (Barlow et al., 2018); (2) to assess the acceptability of the intervention among both recipients and psychotherapists; and (3) to examine preliminary signals of the UP-B's efficacy. The main questions it aims to answer are:

1. Is the intervention feasible as indicated by recruitment rates, data collection procedures, and acceptable rates of participant retention and treatment completion?
2. Is the UP-B acceptable for both participants and psychotherapists considering content, content structure, mode of delivery, and adherence?
3. Does the UP-B show preliminary evidence of effectiveness (i.e., efficacy signals) in reducing burnout, anxiety, depression, and increasing well-being?

DETAILED DESCRIPTION:
This research employs a single-arm, open-label trial design with a one-month follow-up assessment. In addition, two post-intervention focus groups will be conducted-one with participating psychotherapists and one with participants-to explore potential barriers to implementation and to identify the strengths and weaknesses of the intervention.

The Unified Protocol for Burnout consists of eight modules delivered in a group format, with approximately eight participants per group. The intervention is administered across eight two-hour sessions and is designed to treat clinical burnout. Participants will learn a set of transdiagnostic skills aimed at improving their ability to manage burnout and associated symptoms, such as anxiety and depression. These skills include mindful emotion awareness, cognitive flexibility, and strategies for countering maladaptive emotional behaviors.

The psychotherapists involved in the study (n= 3) will receive specialized training in the Unified Protocol and will be supervised throughout the intervention by two licensed clinical psychologists and psychotherapists with extensive experience in developing and implementing the Unified Protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants must score above the moderate burnout threshold on the Burnout Assessment Tool (BAT) to be considered eligible. Those who meet this cutoff will subsequently undergo a structured clinical interview to verify the presence of clinical burnout symptoms. The interview will assess whether the symptom profile is consistent with clinical burnout and will document the onset, progression, and course of symptoms. To be considered eligible for the study, the cause of symptoms must be burnout.

Exclusion Criteria:

* Current engagement in psychotherapy, defined as receiving ongoing psychological treatment at the time of screening;
* Current use of psychotropic medication (e.g., antidepressants, anxiolytics, mood stabilizers);
* Presence of a diagnosed personality disorder and as determined by the clinical interview;
* Presence of a psychiatric disorder;
* Presence or history of a psychotic disorder;
* Suicidal ideation, as assessed through the clinical interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the UP-B | From baseline through post-intervention and 1-month follow-up
  Feasibility will be assessed in terms of recruitment capability, practicality, adaptability, and implementation fidelity. Recruitment capability refers to the number of participants successfully identified and enrolled. Practicality concerns whether the intervention can be delivered using available resources, time, training, and materials. Adaptability refers to the flexibility of the intervention procedures to accommodate diverse needs. Implementation fidelity refers to the extent to which professionals are able to deliver the intervention as intended.
Feasibility: Protocol fidelity (TARS-UP) | From baseline to post-intervention (8 weeks)
  Therapist adherence will be evaluated using the Therapist Adherence Rating Scale for the Unified Protocol (TARS-UP), adapted for use with the Unified Protocol for Burnout. Each intervention module will be evaluated by an observer using a checklist that captures the presence or absence of core treatment components and provides global ratings of therapist performance (e.g., rapport, engagement, session management, and overall session quality).
Module-Specific Acceptability (Participant Perspective) | After each intervention module (across the intervention period)
  A questionnaire assessing participants' module-specific acceptability will be administered following each intervention module. The questionnaire includes five Likert-type items (two assessing group process and three assessing module content) and two open-ended questions designed to capture qualitative feedback.
Module-Specific Acceptability (Psychotherapist Perspective) | After each intervention module (across the intervention period)
  A brief module-specific acceptability questionnaire developed for this study will be administered to psychotherapists following delivery of each intervention module. The questionnaire consists of structured yes/no and yes/somewhat/no questions assessing implementation issues (e.g., barriers to delivery and adequacy of session time), numeric rating questions (1-10) assessing perceived fit of the module content and participant engagement, and open-ended questions allowing therapists to elaborate on their responses and provide feedback on strengths of the module and areas for improvement.
Global Acceptability | Post-intervention (8 weeks)
  An 8-item questionnaire developed by Sekhon et al. (2022) will be used to assess acceptability of the intervention from both participant and psychotherapist perspectives. The questionnaire is based on the Theoretical Framework of Acceptability (TFA). Items corresponding to each TFA construct will be analysed separately. No composite total score will be calculated. Overall acceptability will be assessed using the single general acceptability item.
Behavioral indicators of Acceptability | Post-intervention (8 weeks)
  Attrition will be operationalized in terms of drop-out rates. Adherence will be operationalized as the number of sessions attended and the quality of completed homework assignments.

SECONDARY OUTCOMES:
Burnout | From baseline through post-intervention and 1-month follow-up.
  Burnout will be assessed using the Burnout Assessment Tool-23 (BAT-23; Schaufeli et al., 2020), a 23-item self-report measure rated on a 5-point Likert-type scale. The BAT-23 assesses core burnout symptoms, which can be analysed separately or as a composite score, as well as secondary distress symptoms, which are summed and interpreted as a single score.
Depression Severity | From baseline through post-intervention and 1-month follow-up.
  To assess depression severity, the Overall Depression Severity and Impairment Scale (ODSIS-5; Bentley et al., 2014) will be used. The ODSIS-5 is a 5-item Likert-type scale, with total scores ranging from 0 to 20. Higher scores indicate greater depression severity.
Anxiety Severity | From baseline through post-intervention and 1-month follow-up.
  To assess anxiety severity, the Overall Anxiety Severity and Impairment Scale (OASIS-5; Norman et al., 2006) will be used. The OASIS-5 is a 5-item Likert-type scale, with total scores ranging from 0 to 20. Higher scores indicate greater anxiety severity.
Well-being | From baseline through post-intervention and 1-month follow-up.
  Well-being will be assessed using the The World Health Organization-Five Well-Being Index (WHO-5), a 5-item self-report measure rated on a 6-point Likert-type scale (World Health Organization, Regional Office for Europe, 1998). Total scores range from 0 to 25, with higher scores indicating greater well-being.
Emotion Regulation | From baseline through post-intervention and 1-month follow-up.
  Emotional regulation will be assessed using the Difficulties in Emotional Regulation scale -16 (DERS-16; Bjureberg et al., 2016), an 16-item self-report measure rated on a 5-point Likert scale. Item responses will be summed to yield a total score ranging from 16 to 80, with higher scores indicating greater difficulties in emotion regulation.
Group factors | Post-intervention (8 weeks)
  Group therapeutic processes will be assessed using the Therapeutic Factors Inventory-8 (TFI-8; Tasca et al., 2014), an 8-item self-report measure rated on a 7-point Likert scale. Item responses will be summed to yield a total score ranging from 8 to 56, with higher scores indicating stronger perceived group therapeutic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Rusu, PhD, Principal Investigator — West University of Timisoara
Locations (1):
- West University of Timișoara, Timișoara, Timiș County, Romania

REFERENCES:
- [Background] World Health Organization. Regional Office for Europe; Wellbeing measures in primary health care / the DepCare Project: report on a WHO meeting: Stockholm, Sweden, 12-13 February 1998; World Health Organization. Regional Office for Europe; 1998
- [Background] Bjureberg, J.; Ljótsson, B.; Tull, M. T.; Hedman, E.; Sahlin, H.; Lundh, L.-G.; Bjärehed, J.; DiLillo, D.; Messman-Moore, T.; Gumpert, C. H.; Gratz, K. L.; Development and Validation of a Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16; Journal of Psychopathology and Behavioral Assessment; 2016; 38; 284-296.
- [Background] Bentley, K. H., Gallagher, M. W., Carl, J. R., & Barlow, D. H., Development and validation of the overall depression severity and impairment scale, Psychological assessment, 2014, 26(3), 815.
- [Background] Schaufeli, W. B., De Witte, H. & Desart, S., Manual Burnout Assessment Tool (BAT) - Version 2.0, KU Leuven. 2020, Unpublished internal report.
- [Background] Norman, S. B., Hami Cissell, S., Means-Christensen, A. J., & Stein, M. B., Development and validation of an overall anxiety severity and impairment scale (OASIS), Depression and anxiety, 2006, 23(4), 245-249.
- [Background] Barlow, D. H., Unified protocol for transdiagnostic treatment of emotional disorders: Therapist guide, Oxford University Press, 2018. 2nd edition
- [Background] Tasca, G. A., Cabrera, C., Kristjansson, E., MacNair-Semands, R., Joyce, A. S., & Ogrodniczuk, J. S. The Therapeutic Factors Inventory-8: Using item response theory to create a brief scale for continuous process monitoring for group psychotherapy. 2016. Psychotherapy Research, 26(2), 131-145
- [Background] Tennant, R., Hiller, L., Fishwick, R., Platt, S., Joseph, S., Weich, S., Parkinson, J., Secker, J., & Stewart-Brown, S., The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. 2007. Health and quality of life outcomes, 5, 63.
- [Background] Sekhon, M., Cartwright, M., & Francis, J. J. Development of a theory-informed questionnaire to assess the acceptability of healthcare interventions. BMC health services research, 2022, 22(1), 279.